CLINICAL TRIAL: NCT00089245
Title: Phase I Study Of Intrathecal Radioimmunotherapy Using I-8H9 For Central Nervous System/Leptomeningeal Neoplasms
Brief Title: Radiolabeled MAB Therapy in Patients With Refractory, Recurrent, or Advanced CNS or Leptomeningeal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Corporate business decision. No safety or efficacy concerns.
Sponsor: Y-mAbs Therapeutics (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-133; MSKCC-03133 (Other: Memorial Sloan Kettering Cancer Center)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Brain and Central Nervous System Tumors; Neuroblastoma; Sarcoma
Keywords: leptomeningeal metastases; recurrent neuroblastoma; disseminated neuroblastoma; recurrent adult brain tumor; recurrent childhood medulloblastoma; recurrent childhood rhabdomyosarcoma; recurrent childhood soft tissue sarcoma; recurrent osteosarcoma; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; childhood atypical teratoid/rhabdoid tumor; adult medulloblastoma; previously treated childhood rhabdomyosarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic osteosarcoma; childhood desmoplastic small round cell tumor; metastatic childhood soft tissue sarcoma; adult rhabdomyosarcoma; recurrent adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroblastoma; Sarcoma; Meningeal Carcinomatosis; Brain Neoplasms; Medulloblastoma; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Rhabdoid Tumor; Desmoplastic Small Round Cell Tumor; Rhabdomyosarcoma | interventions — omburtamab I-131

ARMS (1):
- Radiolabeled Monoclonal Antibody Therapy (Experimental): This is a Phase I trial designed to evaluate the Maximally Tolerated Dose (MTD) of intrathecal 131I-8H9. In order to find the MTD, a dose escalation scheme will be employed with patients entering in cohorts of 3 at each dose level from 10 mCi to 60 mCi and a cohort of 6 at each dose level from 70 mCi to 100 mCi.
  Interventions: Drug: Iodine I 131 MOAB 8H9

INTERVENTIONS:
Drug: Iodine I 131 MOAB 8H9 — Patients will be injected, intrathecally, with 2 mCi 131I-Omburtamab during week 1 of a 5 week cycle.
Drug: Iodine I 131 MOAB 8H9 — The dose used in this study is 50 mCi 131IOmburtamab, (averaging 5 mCi/mg Omburtamab at 50 mCi dose) which will be administered to each patient during week 2 of a 5 week cycle.

SUMMARY:
The purpose of this study is to test the feasibility and toxicity of administering intrathecal immunotherapy for patients with central nervous system/leptomeningeal (CNS/LM) malignancies.

DETAILED DESCRIPTION:
This is a phase I study, where the purpose is to find a safe dose of a new medicine called antibody 8H9. Antibodies are made by the body to fight infections and in some cases, to fight tumors. The antibody 8H9 is made by mice and can attack many kinds of tumors. 8H9 antibody can have a dose of radiation attached to it called 131-I. 131I-8H9 has been given in the vein to patients to find cancer cells. This is the first study using 131I-8H9 in the fluid in the spine to kill cancer cells. 131-I is a beta emitting isotope used extensively for radiation targeted therapies.

ELIGIBILITY:
Subject Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of a malignancy known to be 8H9 reactive. 8H9 expression must be confirmed by immunohistochemical staining of tumor and assessed by the Department of Pathology or by immunofluorescence of bone marrow except for patients confirmed to have neuroblastoma.
* Patients must have CNS/ leptomeningeal disease which is refractory to conventional therapies or for which no conventional therapy exists OR a recurrent brain tumors with a predilection for leptomeningeal dissemination (medulloblastoma, PNET, rhabdoid tumor).
* Patients must have no rapidly progressing or deteriorating neurologic examination.
* Patients must have an absolute neutrophil count (ANC) > 1000/ul and a platelet count > 50,000/ul.
* Patients may have active malignancy outside the central nervous system.
* Both pediatric and adult patients of any age are eligible.
* Patients or a legal guardian will sign an informed consent form approved by the IRB and obtained by the Principal or a Co- Investigator before patient entry. Minors will provide assent.
* Patients with stored stem cells will be treated at the escalating dose while patients with no stem cells will be treated at the 50 mCi dose. Neuroblastoma patients can be treated at the 50 mCi dose with or without stored stem cells.

Subject Exclusion Criteria:

* Patients with obstructive or symptomatic communicating hydrocephalus.
* Patients with an uncontrolled life-threatening infection.
* Patients who are pregnant: Pregnant women are excluded for fear of danger to the fetus. Therefore negative pregnancy test is required for all women of child-bearing age, and appropriate contraception is required during the study period.
* Patients who have received cranial or spinal irradiation less than 3 weeks prior to the start of this protocol.
* Patients who have received systemic chemotherapy (corticosteroids not included) less than 3 weeks prior to the start of this protocol.
* Severe major organ toxicity. Specifically, renal, cardiac, hepatic, pulmonary, and gastrointestinal system toxicity should all be less than grade 2. Patients with stable neurological deficits (because of their brain tumor) are not excluded. Patients with <= 3 hearing loss are not excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2004-02-05 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Number of patients that have treatment related toxicities | 2 years
  Assessment of patient with treatment related toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Kim Kramer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Kramer K, Pandit-Taskar N, Kushner BH, Zanzonico P, Humm JL, Tomlinson U, Donzelli M, Wolden SL, Haque S, Dunkel I, Souweidane MM, Greenfield JP, Tickoo S, Lewis JS, Lyashchenko SK, Carrasquillo JA, Chu B, Horan C, Larson SM, Cheung NV, Modak S. Phase 1 study of intraventricular 131I-omburtamab targeting B7H3 (CD276)-expressing CNS malignancies. J Hematol Oncol. 2022 Nov 12;15(1):165. doi: 10.1186/s13045-022-01383-4. PMID 36371226
- [Derived] Yerrabelli RS, He P, Fung EK, Kramer K, Zanzonico PB, Humm JL, Guo H, Pandit-Taskar N, Larson SM, Cheung NV. IntraOmmaya compartmental radioimmunotherapy using 131I-omburtamab-pharmacokinetic modeling to optimize therapeutic index. Eur J Nucl Med Mol Imaging. 2021 Apr;48(4):1166-1177. doi: 10.1007/s00259-020-05050-z. Epub 2020 Oct 13. PMID 33047248
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/